CLINICAL TRIAL: NCT01604057
Title: A Parallel Group Study to Evaluate the Effect of Six Weeks of Treatment With Nasal Spray (NS) ZT-034, Compared to Subcutaneous (SC) Forteo and Placebo, on Bone Formation, as Assessed by Stimulation of Serum P1NP Levels in Postmenopausal Women With Low Bone Mass
Brief Title: Study to Evaluate Effect of Intranasal Teriparatide on Serum P1NP, a Biomarker of Bone Formation, in Postmenopausal Women With Low Bone Mass
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azelon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZT-3201
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Nasal Sprays; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Low Dose Nasal Spray (Experimental)
  Interventions: Drug: ZT-034 Low Dose Nasal Spray
- Mid Dose Nasal Spray (Experimental)
  Interventions: Drug: ZT-034 Mid Dose Nasal Spray
- High Dose Nasal Spray (Experimental)
  Interventions: Drug: ZT-034 High Dose Nasal Spray
- Forteo (Active Comparator): 20ug subcutaneous injection daily
  Interventions: Drug: Teriparatide
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZT-034 Low Dose Nasal Spray — Nasal Spray
  Arms: Low Dose Nasal Spray
Drug: ZT-034 Mid Dose Nasal Spray — Nasal Spray
  Arms: Mid Dose Nasal Spray
Drug: ZT-034 High Dose Nasal Spray — Nasal Spray
  Arms: High Dose Nasal Spray
Drug: Teriparatide — 20 mcg subcutaneous daily
  Other Names: Forteo
  Arms: Forteo
Drug: Placebo — Nasal Spray
  Arms: Placebo Nasal Spray

SUMMARY:
This study is being conducted to evaluate the effect treatment has on serum P1NP levels, a biomarker of bone formation in postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Females Age ≥ 45 years.
* Weight > 45 kg and < 90 kg
* Normal nasal examination at baseline.
* Low bone mass at lumbar spine, total hip or femoral neck (BMD T-score of ≤ - 1.5 or lower) or a recent (within 5 years of baseline) history of fragility fracture (excluding fractures of hands, feet, face and/or skull) and a T-score of -1.0 or lower at lumbar spine, total hip or femoral neck

Exclusion Criteria:

* Serious Medical Condition
* History of diseases which affect bone metabolism other than postmenopausal osteoporosis such as Paget's disease, any secondary causes of osteoporosis, hypoparathyroidism, or hyperparathyroidism
* Have a history of cancer within the past 5 years, except for basal cell carcinoma
* Have hypocalcemia or hypercalcemia from any cause or have a recent history of kidney stones or pre-existing hypercalciuria;
* Have used any of the mostly commonly prescribed osteoporosis medications within 3 months of starting the investigational product, or for more than 1 month at any time within 6 months prior to starting investigational product

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Change in Serum P1NP from baseline to end of treatment. | 6 weeks

SECONDARY OUTCOMES:
Change in serum calcium and incidence of hypercalcemia (pre-dose and post-dose) | baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian MacDonald, Study Director — Azelon Pharmaceuticals